CLINICAL TRIAL: NCT04590183
Title: Peking University Third Hospital Medical Science Research Ethics Committee
Brief Title: The Effectiveness and Safety of FK-506 for the Treatment of Posner-Schlossman Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Chun Zhang, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M2020059
Record Dates: First submitted 2020-09-14; First posted 2020-10-19 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Posner Schlossman Syndrome
Keywords: Posner Schlossman Syndrome; FK-506; effectiveness; safety
MeSH Terms: interventions — Tacrolimus; Pharmaceutical Preparations; prednisolone acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental)
  Interventions: Drug: FK-506 (Drug)
- The control group (Sham Comparator)
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: FK-506 (Drug) — Twice a day
  Other Names: Tacrolimus eye drops
  Arms: The experimental group
Drug: Prednisolone Acetate 1% Oph Susp — Four times a day
  Arms: The control group

SUMMARY:
To evaluate the effectiveness and safety of tacrolimus eye drops (FK-506) in the treatment of Posner-Schlossman Syndrome. It is expected to collect 30 patients with PSS who are in the Ophthalmology Department of Peking University Third Hospital. The included PSS patients were divided into experimental group and control group using simple randomization method. Among them, the experimental group was treated with FK-506 twice a day, and the control group was treated with prednisolone acetate ophthalmic suspension 1% 4 times a day.

For all PSS patients whose intraocular pressure is higher than 30mmHg, also add brinzolamide eye drops 3 times a day. Best corrected visual acuity, Goldmann intraocular pressure, anterior section photographs, corneal endothelial cells，corneal confocal microscope, Heidelberg retinal nerve analysis, Octopus visual field were examined on baseline and 1 week, 2 weeks, 3 weeks, 4 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of PSS Must be able to communicate with doctor and understand this study

Exclusion Criteria:

- Fuchs syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Silt-lamp examination of the cornea | 1 week after the treatment
  KP numbers after the treatment
Silt-lamp examination of the cornea | 2 weeks after the treatment
  KP numbers after the treatment
Silt-lamp examination of the cornea | 3 weeks after the treatment
  KP numbers after the treatment
Silt-lamp examination of the cornea | 4 weeks after the treatment
  KP numbers after the treatment

SECONDARY OUTCOMES:
Goldmann ophthalmotonometer examination of intra-ocular pressure | 1 week after the treatment
  change of intra-ocular pressure
Goldmann ophthalmotonometer examination of intra-ocular pressure | 2 weeks after the treatment
  change of intra-ocular pressure
Goldmann ophthalmotonometer examination of intra-ocular pressure | 3 weeks after the treatment
  change of intra-ocular pressure
Goldmann ophthalmotonometer examination of intra-ocular pressure | 4 weeks after the treatment
  change of intra-ocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chun Zhang, PHD,MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No